CLINICAL TRIAL: NCT07397702
Title: Effects of HIIT and MICT Training on Cardiorespiratory Fitness, Testosterone/Cortisol Ratio, and Mental Health in Young Adults: an 8-week Randomized Clinical Trial
Brief Title: Effects of HIIT and MICT Training on Cardiorespiratory Fitness, Testosterone/Cortisol Ratio, and Mental Health in Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Colima (Other)
Responsible Party: Principal Investigator, Pedro Julian Flores Moreno, Ph. D. in Science, Universidad de Colima
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2025-23b
Record Dates: First submitted 2026-01-05; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Exercise
Keywords: High-Intensity Interval Training; Aerobic Exercise; Testosterone; Cortisol; Anxiety Disorders; Depressive Disorder
MeSH Terms: conditions — Motor Activity; Anxiety Disorders; Depressive Disorder | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Beck scales will be applied to assess anxiety and depression. Subsequently, cardiorespiratory fitness will be assessed by means of the Course Navette test, which consists of running at a progressive speed in 20 meters delimited following a sound signal until exhaustion, at the end of the test the final distance run is recorded and converted into VO2max. These measurements will be performed during week 0 (pre-training) and week 8 (post-training). Training intensity will be monitored by maximum heart rate (HRmax), using Polar H10 heart monitors, and will be complemented with the subjective perception of exertion scale, following the recommendations of the American College of Sports Medicine. Training programs: a) HIIT group: running 10 repetitions of 1-minute intervals at 85-90% of HRmax, interspersed with 1-minute recovery at 50-60% of HRmax. b) MICT group: perform 30 minutes of continuous aerobic running at 60-70% of HRmax, with a frequency of 3 weekly sessions.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: high-intensity interval training program (Experimental): High-intensity interval training (HIIT) sessions will consist of continuous running for a 5-minute warm-up at 75% of maximum heart rate (HRmax), followed by 10 repetitions of intermittent running in 1-minute intervals at 85-90% of HRmax, intercalated with 1-minute recovery periods at 50-60% of HRmax. There will be 3 sessions per week (75-minute weekly training). All HIIT intervention sessions end with a cool-down walk and stretching.
  Interventions: Other: High-intensity interval training
- Group B: moderate-intensity continuous training program (Active Comparator): Moderate-intensity continuous training (MICT) sessions will consist of running continuously for 30 minutes at an intensity of 60-70% of HRmax, with a frequency of 3 sessions per week (60 minutes of training per week). All sessions with MICT intervention end with a cool-down walk and stretching.
  Interventions: Other: Moderate-intensity continuous training

INTERVENTIONS:
Other: High-intensity interval training — The intervention involves physical exercise with the aim of observing any changes that may occur in mental health and hormonal parameters. However, the magnitude of these effects and the type of exercise that is most effective in reducing symptoms of anxiety and depression are still unknown.
  Arms: Group A: high-intensity interval training program
Other: Moderate-intensity continuous training — The intervention involves physical exercise with the aim of observing any changes that may occur in mental health and hormonal parameters. However, the magnitude of these effects and the type of exercise that is most effective in reducing symptoms of anxiety and depression are still unknown.
  Arms: Group B: moderate-intensity continuous training program

SUMMARY:
This study will use a randomized, double-blind clinical trial to evaluate the effects of eight-week HIIT and MICT exercise programs on cardiorespiratory fitness, the testosterone/cortisol ratio, and mental health in 68 healthy, moderately active young adults aged 18 to 21. Participants will be assigned to parallel groups based on their sex and training type (HIIT men, HIIT women, MICT men, MICT women). The key metrics will be measured both before and after the intervention period to assess the impact of the different training regimens.

DETAILED DESCRIPTION:
This randomized, double-blind clinical trial will investigate the effects of high-intensity interval training (HIIT) versus moderate-intensity continuous training (MICT) on cardiorespiratory fitness and symptoms of anxiety and depression in high school students.

The study will recruit 68 male and female students, aged 15-19, who are moderately inactive. Participants will be randomized into HIIT or MICT groups, stratified by gender. The 8-week intervention consists of three weekly sessions: HIIT involves 10x1-minute high-intensity intervals, while MICT consists of 30 minutes of continuous running. Cardiorespiratory fitness (measured via the Course Navette test to estimate VO₂max) and mental health symptoms (using Beck inventories) will be assessed before and after the intervention.

The primary hypothesis is that HIIT will yield greater improvements in VO₂max and greater reductions in anxiety and depression symptoms compared to MICT. Statistical analysis will employ ANOVA and related tests to evaluate changes within and between groups, with a significance level set at p<0.05. The study aims to provide evidence for designing personalized exercise programs that optimize both physical and mental health in adolescents.

ELIGIBILITY:
Inclusion criteria:

* Men and women aged 18 to 21.
* Lead a sedentary or moderately active lifestyle (IPAQ ≤600 METs-min/week).
* Subjects diagnosed by a physician as fit for physical exercise.
* Informed consent form signed by the study subjects.

Exclusion criteria:

* Subjects with any motor disability.
* Pregnant women.
* Subjects with metabolic disorders.
* Subjects with chronic respiratory diseases such as asthma, emphysema, or cancer, obstructive pulmonary disease.
* Subjects with high blood pressure or arrhythmia.
* Failure to sign the informed consent form.
* Subjects who are in a high-performance physical training program.
* Women with irregular menstrual cycles who take contraceptive medication to regulate their menstrual cycle.
* Consumption of caffeine, alcohol, and tobacco or use of electronic cigarettes.
* Subjects with a cyclical diagnosis of anxiety and depression by a specialist.
* Frequent consumption of alcoholic beverages (more than 7 drinks per week for women and more than 14 drinks per week for men) or a history of excessive alcohol consumption.
* Subjects who consume dietary supplements (caffeine, nitric oxide precursors, beta-alanine, creatine, sodium bicarbonate, or L-carnitine).

Elimination criteria:

* Voluntary withdrawal from the study.
* Attendance at less than 80% of intervention sessions.
* Incomplete measurement schedule or insufficient sample size.
* Joint or muscle injuries caused by the training program.
* Overtraining syndrome.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-05-25 (Estimated); Primary Completion 2026-07-24 (Estimated); Study Completion 2026-08-07 (Estimated)

PRIMARY OUTCOMES:
Symptoms of anxiety from baseline to eight weeks. | Baseline and week 8 of training.
  The measurement of anxiety symptoms will be conducted using the Beck Anxiety Inventory (BAI) in printed format, which is a validated psychological tool used to assess the severity of anxiety symptoms in adults. The total score is interpreted on a scale from 0 to 63, where a score of 0 indicates the absence of anxiety symptoms, and higher scores reflect increasing levels of anxiety, with the upper values representing severe anxiety.
Symptoms of depression from baseline to eight weeks. | Baseline and week 8 of training.
  The measurement of depression symptoms will be conducted using the Beck Depression Inventory (BDI) in printed format, which is a validated psychological tool used to assess the severity of depression symptoms in adults. The total score is interpreted on a scale from 0 to 63, where a score of 0 indicates the absence of depression symptoms, and higher scores reflect increasing levels of depression, with the upper values representing severe depression.
Testosterone levels using the ELISA method | Baseline and week 8 of training.
  Testosterone and cortisol levels will also be determined in picograms per milliliter (pg/mL) using the enzyme-linked immunosorbent assay (ELISA) method, which is employed to quantify hormones, cytokines, and other proteins in blood or other biological fluids.
Cortisol levels using the ELISA method | Baseline and week 8 of training.
  Cortisol levels will also be determined in picograms per milliliter (pg/mL) using the enzyme-linked immunosorbent assay (ELISA) method, which is employed to quantify hormones, cytokines, and other proteins in blood or other biological fluids.
Cardiorespiratory capacity using VO₂max | Baseline and week 8 of training.
  Cardiorespiratory capacity will be assessed using the 20-meter run test, with maximal oxygen uptake (VO₂max), expressed in millilitres per minute per kilogram (mL/kg/min), as the main indicator. The test consists of running back and forth between two points separated by 20 meters, following a pace dictated by auditory signals; as the test progresses, the running speed gradually increases.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Julián Flores Moreno, Study Chair — Universidad de Colima

IPD SHARING:
Plan to Share IPD: Yes
the plan to share information with other researchers through the publication of different articles that can be extracted from the research
Supporting Information: Study Protocol, ICF
Time Frame: The information will be available as of August 2026
Access Criteria: To have access to these data, other researchers must be performing the same methodological design, so there is no point in sharing it with a different study design

REFERENCES:
- [Result] Velasco-Orjuela GP, Dominguez-Sanchez MA, Hernandez E, Correa-Bautista JE, Triana-Reina HR, Garcia-Hermoso A, Pena-Ibagon JC, Izquierdo M, Cadore EL, Hackney AC, Ramirez-Velez R. Acute effects of high-intensity interval, resistance or combined exercise protocols on testosterone - cortisol responses in inactive overweight individuals. Physiol Behav. 2018 Oct 1;194:401-409. doi: 10.1016/j.physbeh.2018.06.034. Epub 2018 Jun 22. PMID 29940266
- [Result] Paolucci EM, Loukov D, Bowdish DME, Heisz JJ. Exercise reduces depression and inflammation but intensity matters. Biol Psychol. 2018 Mar;133:79-84. doi: 10.1016/j.biopsycho.2018.01.015. Epub 2018 Feb 3. PMID 29408464
- See also: Transforming mental health for all — https://www.who.int/teams/mental-health-and-substance-use/world-mental-health-report